CLINICAL TRIAL: NCT05644379
Title: An Open, Single-arm, Single-centre Clinical Study Evaluating Cadonilimab Injection in Combination With Regorafenib for the Treatment of Intermediate to Advanced Hepatocellular Carcinoma That Has Failed at Least One Prior Systemic Therapy
Brief Title: A Study Evaluating Cadonilimab Injection in Combination With Regorafenib for the Advanced Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-C-N1-0004
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced Hepatocellular Carcinoma That Has Failed at Least One Prior Systemic Therapy
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab Injection in combination with Regorafenib (Experimental): Cadonilimab Injection in combination with Regorafenib
  Interventions: Drug: Cadonilimab Injection; Drug: Regorafenib

INTERVENTIONS:
Drug: Cadonilimab Injection — Cadonilimab Injection, 6mg/kg, intravenous drip ,q2w,
  Other Names: AK104
Drug: Regorafenib — Regorafenib 80mg, po, orally once daily

SUMMARY:
To evaluate the efficacy and safety of Cadonilimab Injection in combination with Regorafenib in the treatment of intermediate to advanced hepatocellular carcinoma that has failed at least one prior systemic therapy .

DETAILED DESCRIPTION:
An open, single-arm, single-centre clinical study evaluating Cadonilimab Injection in combination with Regorafenib for the treatment of intermediate to advanced hepatocellular carcinoma that has failed at least one prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent signed prior to enrolment.
2. age > 18 years, both sexes
3. patients with histologically or pathologically confirmed intermediate to advanced hepatocellular carcinoma.
4. intermediate to advanced HCC previously treated with anti-PD-1/PD-L1 combined with anti-vascular targeting agents for HCC, with disease progression.
5. Child-Pugh A or B.
6. with measurable lesions (≥10 mm long diameter on CT scan for non-lymph node lesions and ≥15 mm short diameter on CT scan for lymph node lesions according to RECIST 1.1 criteria).
7. ECOG PS score: 0 to 1.
8. expected survival of >12 weeks.
9. function of vital organs in accordance with the following requirements (excluding the use of any blood components and cell growth factors within 14 days).

1) Blood count. Neutrophils ≥ 1.5 x 109/L Platelet count ≥ 60×109/L haemoglobin ≥ 90 g/L. 2) Liver and kidney function. Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula).

total bilirubin (TBIL) ≤ 3 times the upper limit of normal (ULN) Glutamic aminotransferase (AST) or glutamic aminotransferase (ALT) levels ≤ 10 times the upper limit of normal (ULN); urine protein < 2+; if urine protein ≥ 2+, 24-hour urine protein quantification must show ≤ 1 g of protein.

10. normal coagulation function, no active bleeding or thrombotic disease

1. International normalised ratio INR ≤ 1.5 x ULN.
2. partial thromboplastin time APTT ≤ 1.5 x ULN.
3. prothrombin time PT ≤ 1.5 x ULN. 11. Female patients who are non-surgically sterilised or of childbearing age are required to use a medically approved contraceptive (e.g. IUD, pill or condom) during and for 3 months after the end of the study treatment period; female patients of childbearing age who are non-surgically sterilised must have a negative serum or urine HCG test within 7 days prior to study entry; and must be non-lactating; male patients who are non-surgically sterilised or of childbearing age Patients, need to agree to use a medically approved form of contraception with their spouse during and for 3 months after the end of the study treatment period.

12. The subject is voluntarily enrolled in the study, is compliant and cooperates with safety and survival follow-up Exclusion criteria： Exclusion criteria Patients with any of the following are not eligible for enrollment in this study.

1. Subjects with previous or concurrent other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix).
2. the subject has received previous immunotherapy other than anti-PD-1/PD-L1 monoclonal antibody; the subject is known to have a previous allergy to macromolecular protein agents, or is known to be allergic to the components of the drug applied.
3. The subject has any active autoimmune disease or history of autoimmune disease (e.g. the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enterocolitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, previous thyroid surgery cannot be included; the subject has vitiligo or has complete remission of asthma in childhood and in adulthood (subjects who do not require any intervention can be included; subjects with asthma requiring medical intervention with bronchodilators cannot be included).
4. subjects who are on immunosuppressive, or systemic, or absorbable topical hormone therapy for immunosuppressive purposes (doses >10 mg/day of prednisone or other isotonic hormones) and who continue to use them within 2 weeks prior to enrolment
5. have clinically symptomatic ascites or pleural effusion requiring therapeutic puncture or requiring frequent drainage of ascites (≥1 time/month)
6. subjects with clinically symptomatic cardiac conditions or diseases that are not well controlled, such as (1) NYHA class 2 or higher heart failure (2) unstable angina pectoris (3) previous myocardial infarction within 1 year (4) patients with clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention
7. subjects with active infection or unexplained fever >38.5 degrees during screening and prior to the first dose (subjects with fever arising from a tumour may be enrolled, as judged by the investigator)
8. patients with previous and current objective evidence of a history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, or severely impaired lung function
9. subjects with congenital or acquired immune deficiency, e.g. HIV infection
10. subjects who have received a live vaccine less than 4 weeks prior to study drug administration or possibly during the study period
11. subjects with a known history of psychotropic substance abuse, alcoholism or drug use
12. patients who are unable to administer the drug orally
13. have received herbal or proprietary Chinese medicine with an anti-tumour indication within 2 weeks prior to the first dose .

14 Patients who, in the opinion of the investigator, should be excluded from the study, for example, subjects who, in the judgment of the investigator, have other factors that may force the study to be terminated, e.g., other serious illnesses (including psychiatric illnesses) requiring comorbid treatment, severe fundic esophageal varices, serious laboratory test abnormalities, accompanying family or social factors that would compromise the safety of the subject, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Overall response rate ( ORR) | up to 1 years
  Defined as proportion of patients who have a best response of CR or PR
Overall survival (OS) | up to 3 years
  OS is defined as the time from date of neoadjuvant treatment start to the date of death from any cause or to the date of last follow-up if patients are alive. If a patient is alive by the time of final analysis, the patient will be censored at the last follow-up date.
Progress Free Survival （PFS） | up to 3 years
  Defined as the time from enrollment to disease progression or death (whichever occurs first)
Adverse Events (AEs) | up to 3 years
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No